CLINICAL TRIAL: NCT01247870
Title: A Randomised, Double-blind, Placebo-controlled Trial of Metformin in Chronic Obstructive Pulmonary Disease (COPD) Exacerbations: a Pilot Study
Brief Title: Metformin in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: St George's, University of London (Other)
Collaborators: Medical Research Council (Other Government); British Lung Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10.0086; 2010-020818-28 (EudraCT Number)
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease, COPD, metformin
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Metformin (Experimental): Metformin 1 g twice daily for 28-35 days
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Matched placebo capsules
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin 1 g twice daily for 28-35 days
  Arms: Metformin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effect of a tablet medication, called metformin, in flare-ups (exacerbations) of chronic obstructive pulmonary disease. The investigators believe that metformin may effectively control the blood sugar level during COPD exacerbations. This is important because there is evidence that a high blood sugar level during exacerbations may be linked with a worse prognosis. The investigators also think that metformin may have other potentially useful effects on inflammation, antioxidant levels, the effectiveness of steroid treatment, and recovery.

DETAILED DESCRIPTION:
Does metformin lower the blood sugar level in patients suffering from exacerbations of chronic obstructive pulmonary disease (COPD)?

COPD is the fourth leading cause of death worldwide, and a major cause of ill health. In the UK, it affects some 3.7 million people and causes over 30,000 deaths per year. It is usually, but not always, caused by smoking. Most people affected are over 65-years-old. Sufferers experience progressively worsening cough, sputum production, breathlessness and exercise limitation. This is punctuated by 'flare-ups' (exacerbations), when their symptoms worsen substantially. Approximately 25% of patients hospitalised for exacerbations die within a year, and over 50% within 5 years. There is a pressing need for new and improved treatments for COPD exacerbations.

This study will assess the effect of metformin, a tablet medication, in COPD exacerbations. Metformin has been in common use for over 50 years in patients with diabetes, to lower the blood sugar level. In COPD exacerbations, the blood sugar level is often high, and the higher it is, the more likely the patient will have a poor outcome. This led us to speculate that lowering the sugar level with metformin may improve outcomes from COPD exacerbations. However, COPD and diabetes are quite different diseases, and the investigators do not know whether metformin will work as a sugar-lowering medicine in COPD exacerbations. The investigators need to confirm this before the investigators can perform larger studies to assess its effect on outcomes such as readmission and mortality rates.

The investigators will test this medicine in a 1-month trial in patients hospitalised for COPD exacerbations. The target sample size is 69 patients, with a minimum of 48 patients required for primary endpoint analysis. Two-thirds of the patients will take metformin, and one-third a dummy (placebo) tablet. Neither the patients nor the researchers know who is taking which. The investigators will measure their sugar levels by regular finger-prick tests, and then compare the average readings in the two groups. The investigators will also assess the medicine's effects on other markers of blood sugar level, and carry out additional exploratory investigations on the effect of the medicine on clinical outcomes, markers of inflammation, and markers of oxidative/carbonyl stress and steroid responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD
* Hospitalisation for exacerbation of COPD
* Age ≥35 years
* Expected to remain in hospital for at least 48 hours

Exclusion Criteria:

* Prior diagnosis of diabetes mellitus requiring insulin or oral hypoglycaemic therapy
* Hypersensitivity to metformin hydrochloride or to any of the excipients
* Renal impairment
* Severe sepsis
* Metabolic acidosis
* Decompensated type 2 respiratory failure
* Severe congestive cardiac failure
* Acute coronary syndrome
* Hepatic insufficiency
* Excessive alcohol consumption
* Malnourished or at high risk for malnutrition
* Moribund or not for active treatment
* Admitted to critical care unit
* Unable to give informed consent
* Pregnancy or lactation

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-01; Primary Completion 2014-03 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Capillary glucose concentration | During hospitalisation period
  The mean capillary glucose concentration during hospitalisation period following study entry, as a measure of both efficacy and safety.

SECONDARY OUTCOMES:
COPD Assessment Test score | Study entry, hospital discharge, and follow-up
Exacerbation of Chronic Pulmonary Disease Tool (EXACT) score | Days 5, 10 and 28
Time to discharge | Hospital discharge
  Number of days from hospital admission to hospital discharge
Recurrent exacerbation, readmission, and death rate | 3 months
  Rates of recurrent exacerbation (defined as treatment with antibiotics and/or systemic corticosteroids for breathlessness, cough or wheeze), readmission to hospital, or death
Insulin requirement during hospitalisation period | During hospitalisation period following study entry
  Mean daily insulin use during hospitalisation period following study entry
Haemoglobin A1c | Follow-up (one month post study entry)
  Mean haemoglobin A1c concentration
C-reactive protein concentration | Days 7 and follow-up (one month)
  Mean concentration of C-reactive protein in the blood
Body mass index | Follow-up (one month)
Waist circumference | Follow-up (one month)
Forced expiratory volume in 1 second | At hospital discharge and follow-up (one month)
  Mean forced expiratory volume in 1 second (FEV1) expressed as a percentage of predicted value
Fructosamine | At hospital discharge and follow-up (one month)
  Mean serum fructosamine concentration
Interleukin 6 | At hospital discharge and follow-up (one month)
  Serum concentration of IL-6 (absolute value and change from baseline)
Interleukin 8 | At hospital discharge and follow-up (one month)
  Serum concentration of IL-8 (absolute value and change from baseline)
Tumor necrosis factor alpha | At hospital discharge and follow-up (one month)
  Serum concentration of TNF-alpha (absolute value and change from baseline)
Interferon gamma | At hospital discharge and follow-up (one month)
  Serum concentration of IFN-gamma (absolute value and change from baseline)
8-isoprostane | At hospital discharge and follow-up (one month)
  Serum concentration of 8-isoprostane (absolute value and change from baseline)
Total carbonyl stress | At hospital discharge and follow-up (one month)
  Total carbonyl stress, measured in serum (absolute value and change from baseline)
Glutathione reduced vs oxidised | At hospital discharge and follow-up (one month)
  Glutathione reduced vs oxidised, measured in serum (absolute value and change from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Emma H Baker, MBChB PhD, Study Chair — St George's, University of London; Andrew W Hitchings, BSc MBBS, Principal Investigator — St George's Healthcare NHS Trust
Locations (9):
- United Kingdom (9):
  - North Tees and Hartlepool NHS Trust, Hartlepool, Cleveland
  - University Hospitals of Morecambe Bay NHS Trust, Lancaster, Cumbria
  - East Sussex Healthcare NHS Trust, Hastings, East Sussex
  - Blackpool Teaching Hospitals NHS Trust, Blackpool, Lancashire
  - Lancashire Teaching Hospitals NHS Trust, Preston, Lancashire
  - Sherwood Forest Hospitals NHS Trust, Sutton in Ashfield, Nottinghamshire
  - Chelsea and Westminster Hospital, London
  - St George's Hospital, London
  - Freeman Hospital, Newcastle

REFERENCES:
- [Derived] Hitchings AW, Baker EH, Jones PW. Handling missing items in the Exacerbations of Chronic Pulmonary Disease Tool. Eur Respir J. 2016 Aug;48(2):564-6. doi: 10.1183/13993003.00269-2016. Epub 2016 May 12. No abstract available. PMID 27174882
- [Derived] Hitchings AW, Lai D, Jones PW, Baker EH; Metformin in COPD Trial Team. Metformin in severe exacerbations of chronic obstructive pulmonary disease: a randomised controlled trial. Thorax. 2016 Jul;71(7):587-93. doi: 10.1136/thoraxjnl-2015-208035. Epub 2016 Feb 25. PMID 26917577